CLINICAL TRIAL: NCT06160154
Title: Minimally Invasive Robot-assisted and Laparoscopic Distal Pancreatectomy in a Pan-European Registry
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M.G. Besselink, Professor of HPB Surgery, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NP5627
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Pancreas Disease
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — all patients undergoing minimally invasive distal pancreatectomy, no intervention, no randomization

SUMMARY:
A planned analysis of outcomes among consecutive patients after MIDP from centers participating in the E-MIPS registry (2019-2021). Main outcomes of interest were intraoperative events, major morbidity (Clavien-Dindo grade ≥3) and 30-day/in-hospital mortality.

DETAILED DESCRIPTION:
The European registry for Minimally Invasive Pancreatic Surgery (E-MIPS) is an E-AHPBA endorsed registry with the aim to monitor and safeguard the introduction of MIPS in Europe. International multicenter audit-based studies focusing on outcomes of minimally invasive distal pancreatectomy (MIDP) are lacking.

A planned analysis of outcomes among consecutive patients after MIDP from centers participating in the E-MIPS registry (2019-2021). Main outcomes of interest were intraoperative events, major morbidity (Clavien-Dindo grade ≥3) and 30-day/in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

Data from all patients who underwent laparoscopic or robotic distal pancreatecromy between January 1st 2019 and December 31st 2021 were included

Exclusion Criteria:

Other pancreatic procedures Hybrid approaches (reconstruction phase open) Procedures with insufficient baseline data / missing primary outcome data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent laparoscopic or robotic distal pancreatecromy between January 1st 2019 and December 31st 2021
Sampling Method: Non-Probability Sample
Enrollment: 1672 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative events | 30 days
  Major bleeding or change in operation
30-day/in-hospital mortality. | 30 days
  Dead in hospital or within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, locatie AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Bodegraven EA, van Ramshorst TME, Bratlie SO, Kokkola A, Sparrelid E, Bjornsson B, Kleive D, Burgdorf SK, Dokmak S, Groot Koerkamp B, Cabus SS, Molenaar IQ, Boggi U, Busch OR, Petric M, Roeyen G, Hackert T, Lips DJ, D'Hondt M, Coolsen MME, Ferrari G, Tingstedt B, Serrablo A, Gaujoux S, Ramera M, Khatkov I, Ausania F, Souche R, Festen S, Berrevoet F, Keck T, Sutcliffe RP, Pando E, de Wilde RF, Aussilhou B, Krohn PS, Edwin B, Sandstrom P, Gilg S, Seppanen H, Vilhav C, Abu Hilal M, Besselink MG; European Consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). Minimally invasive robot-assisted and laparoscopic distal pancreatectomy in a pan-European registry a retrospective cohort study. Int J Surg. 2024 Jun 1;110(6):3554-3561. doi: 10.1097/JS9.0000000000001315. PMID 38498397